CLINICAL TRIAL: NCT01571700
Title: Investigation of Dysynchrony in Patients With Pulmonary Hypertension
Status: Enrolling by invitation | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey A. Feinstein, Principle Investigator, Stanford University
Other Study IDs: DS6901
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Hypertension
Keywords: Mechanical Dysynchrony; Electrical Dysynchrony
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study: Patients with pulmonary hypertension.
  Interventions: Procedure: Catheterization Pacing
- Control: ASD patients or patients with normal hearts

INTERVENTIONS:
Procedure: Catheterization Pacing — The second part of the study will include patients with pulmonary hypertension >5 who are scheduled for a cardiac catheterization for clinical reasons. We will at the conclusion of the routine catheterization, place two pacing catheters within the right atrium and right ventricle and pace the heart at a rate approximately 10% higher than sinus rhythm for 5 minutes. We will then measure dP/dT max in the ventricles, blood pressure and cardiac output using a Fick equation to assess hemodynamics. We will repeat this 3 times using different sites in the right ventricle while simultaneously obtaining echoes to assess mechanical synchrony.
  Groups: Study

SUMMARY:
The purpose of the study is to determine whether patients with pulmonary hypertension (PH) have dysynchrony, and if so whether it is electrical or mechanical. Once this has been determined, during a catheterization the investigators will test if pacing the heart improves blood circulation.

DETAILED DESCRIPTION:
This is a two part study of ventricular dysynchrony in patients with pulmonary hypertension. The first part is an observational study, reviewing routinely obtained clinical information (such as echocardiograms) to assess whether patients with pulmonary hypertension have electrical or mechanical dysynchrony. If so, we will proceed to the second part of the study which will assess whether temporarily pacing the right ventricle, during a clinically indicated catheterization can acutely improve hemodynamics. We will also gather control data for phase 1 from clinically indicated echos and ECG's in patients with ASD's (RV volume load) and in patients who are evaluated for an innocent murmur ( Nl heart). We hope to learn whether patients with pulmonary hypertension, and compromised right ventricles have electrical and mechanical dysnchrony. If this is true, it is theoretically possible that resynchronization (pacing) of the right ventricle could improve hemodynamics, symptoms and long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary artery mean pressure at rest of 25 mm Hg
* Controls (for phase 2) Patients undergoing transcatheter closure of secundum ASD Patients undergoing echocardiogram and ECG as part of work-up for functional murmur who have normal intracardiac anatomy

Exclusion Criteria:

* Reversible cause of pulmonary hypertension
* Age < 5 yrs (for phase 2)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be approached during their routine pulmonary hypertension clinic visit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-09; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Electrical or Mechanical Dysynchrony | Open

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Feinstein, MD, MPH, Principal Investigator — Stan
Locations (1):
- Stanford Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication